CLINICAL TRIAL: NCT03469466
Title: Remotely Guided Ultrasound Among Non-Medical Personnel To Assess Normal Lung Parenchyma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Sahar Ahmad, Assistant Professor, Department of Medicine, Stony Brook University
Other Study IDs: 1190543-1
Record Dates: First submitted 2018-02-13; First posted 2018-03-19 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- untrained: Volunteers untrained in bedside ultrasound technique
- trained: Volunteers previously trained and experienced in bedside ultrasound technique
- healthy volunteer: Standardized patient who will undergo ultrasound study
  Interventions: Diagnostic Test: bedside ultrasound

INTERVENTIONS:
Diagnostic Test: bedside ultrasound — bedside ultrasound imaging of the lungs
  Groups: healthy volunteer

SUMMARY:
This study will assess the feasibility of remotely guided US use by individuals without ultrasound training to assess for normal lung parenchyma in healthy volunteers. The untrained operators (operators) will perform US examinations of lung under the guidance of a medical professional (professional) with experience in ultrasound technique. The professional will guide the operator step by step on how to conduct an US exam of the 'patient's' lung. Images will then be saved and reviewed at a later time by an ultrasound expert to determine quality and clinical functionality in recognizing normal lung parenchyma. This simulation will be analogous to an untrained US operator assessing a potentially ill patient with the assistance of a remotely located physician. An example of this would be an astronaut with respiratory distress after experiencing a rapid decompression event being evaluated by another healthy astronaut by US under the guidance of the flight surgeon at Mission Control.

DETAILED DESCRIPTION:
Volunteers will meet with study personnel in the Clinical Skills Center at Stonybrook University. Informed consent will be obtained from all groups ('operators', 'patients', 'clinicians'). A survey will be conducted to evaluate the subjects' prior experience in ultrasound. Subjects who qualify will continue to participate in the study.

The 'patient' will initially be evaluated by US by an expert and 'ideal' images will be captured and stored for later comparison against those obtained by 'operators'.

The 'operator' will be given an smart phone/table with video communication function and will be connected with the US 'expert', who will be located in a different room, physically and audibly out of range. For the first portion of the study, the 'expert' will instruct the 'operator' on how to conduct an US exam limited to the lung. Using the two-way video and audio communication through the video communication application, the expert will guide to the operator on how to utilize the US machine, where to place the probe, and how to capture and save images. The 'patient' will be instructed not to assist the 'operator' in any way. For the second portion of the study, the 'operator' will utilize the US machine to conduct a similarly limited lung exam on themselves, again with the assistance of the 'expert' but no other study personnel.

Finally, the 'clinicians' will carry out similarly limited lung exams on the 'patient', first without instruction from the 'expert' and then again under similar guidance as the previous portions of the study.

During all portions of the study, time to image capture will be measured by observing personnel. All captured images will be sent to expert reviewers at which time a quality score will be generated. The score will be generated based off of the clinical utility of the image, general image quality, and several technical components of the image. Please see the accompanying Score Sheet for further details. Reviewers will be blinded as to the origin of the images ('operator' vs. 'clinician'). Scores obtained from 'operators' will be compared against those of 'clinicians'. Reviewers will be comprised of three experts in the field of US, all MDs who have received formal training in US and have at least 5 years of clinical US practice experience. Each captured image will be reviewed and scored by all three reviewers.

ELIGIBILITY:
Inclusion Criteria:

* agreeable to consent

Exclusion Criteria:

* refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers agreeable to consent to study and perform bedside ultrasound imaging
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Image Quality | 1 day
  Ultrasound experts will blindly evaluate images obtained from both untrained and trained groups. Using the 'Ultrasound Quality Scorecard', evaluators will assess the quality of the image obtained and the technique carried out to obtain the image. These quality and technique criteria include 'Discernable Lung Parenchyma', 'Presence of A-lines', 'Lack of Obstruction from Rib Shadowing', 'Correct Probe Selection', Correct Depth Setting', 'Correct Gain Selection'. For each criterion (both quality and technique), a binary 'Yes/No' score will be given. Total 'Yes' scores will be summed for each ultrasound exam (minimum 0, maximum 6), with the higher number of 'Yes' responses signifying a higher quality ultrasound exam. Each ultrasound exam will be scored by three separate experts, with the average of the three scores being reported as the 'final score'.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Ahmad, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wimalasena Y, Windsor J, Edsell M. Using ultrasound lung comets in the diagnosis of high altitude pulmonary edema: fact or fiction? Wilderness Environ Med. 2013 Jun;24(2):159-64. doi: 10.1016/j.wem.2012.10.005. Epub 2013 Feb 28. PMID 23453728
- [Result] Lerner DJ, Parmet AJ, Don S, Shimony JS, Goyal MS. Technique for Performing Lumbar Puncture in Microgravity Using Portable Radiography. Aerosp Med Hum Perform. 2016 Aug;87(8):745-7. doi: 10.3357/AMHP.4601.2016. PMID 27634611
- [Result] Martin DS, Caine TL, Matz T, Lee SM, Stenger MB, Sargsyan AE, Platts SH. Virtual guidance as a tool to obtain diagnostic ultrasound for spaceflight and remote environments. Aviat Space Environ Med. 2012 Oct;83(10):995-1000. doi: 10.3357/asem.3279.2012. PMID 23066623
- [Result] Galdamez LA, Clark JB, Antonsen EL. Point-of-Care Ultrasound Utility and Potential for High Altitude Crew Recovery Missions. Aerosp Med Hum Perform. 2017 Feb 1;88(2):128-136. doi: 10.3357/AMHP.4640.2017. PMID 28095957

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT03469466/Prot_SAP_000.pdf